CLINICAL TRIAL: NCT04373473
Title: A Phase 2a, Randomized, Double-blinded, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Lyophilized Fecal Microbiota Transplantation (PRIM-DJ2727) Administered Orally in Combination With Standard of Care Therapy for Prevention of Relapse or Intestinal Inflammation in Adults With Ulcerative Colitis
Brief Title: Evaluation the Safety and Efficacy of Lyophilized Fecal Microbiota Transplantation Administered Orally for Prevention of Relapse or Intestinal Inflammation in Adults With Ulcerative Colitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Herbert DuPont, MD, Professor of Infectious Diseases, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-20-0316
Expanded Access: NCT03786900 (Available)
Record Dates: First submitted 2020-04-28; First posted 2020-05-04 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Adults With Ulcerative Colitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with UC will receive FMT capsules (Experimental): Patients with ulcerative colitis will receive fecal microbiota capsules from 3 healthy donors
  Interventions: Drug: PRIM-DJ2727
- Patients with UC will receive placebo (Placebo Comparator): Patients with ulcerative colitis will receive matching placebo capsules. Placebo capsule will be identical to PRIM-DJ2727 but will not contain intestinal bacteria.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: PRIM-DJ2727 — Fecal Microbiota Transplantation (FMT) product manufactured as PRIM-DJ2727 capsules consists of lyophilized microbiota suspension from well-screened donors. Microbiota from three donors will be combined to make the product.
  Arms: Patients with UC will receive FMT capsules
Drug: Placebos — Placebo capsule will be identical to PRIM-DJ2727 but will not contain intestinal bacteria.
  Arms: Patients with UC will receive placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of lyophilized PRIM-DJ2727 capsules given orally in subjects with ulcerative colitis at remission stage. This study will also include longitudinal analyses of recipient's gut microbiota taxonomy and metagenomics to determine potential associations with clinical outcomes in context of active FMT or placebo administration.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥18 years of age
2. History of active UC in the past 12 months based on standard clinical, endoscopic, or histologic criteria.
3. Remission of UC based on clinical grounds (partial Mayo score of ≤2 with each subscore ≤1), and on stable maintenance therapy.
4. Sexually active male and female subjects of childbearing potential must agree to use an effective method of birth control during the study.
5. Female subjects of childbearing potential must have a negative urine Qualitative HCG pregnancy test at enrolment and on the Week 1, Day 1 of the Treatment prior to administration of study drug.
6. Willing and able to sign an informed consent form and attend all study-related clinic visits, assessments, and follow-up phone calls.
7. Subject has an attending physician who will provide the non-FMT care.

Exclusion Criteria:

1. Unable to take multiple capsules orally.
2. Females who are pregnant, breastfeeding, or planning to become pregnant during the study.
3. Receipt of systemic non-topical antibiotics within 14 days of treatment day 1.
4. Positive results for active HIV, Hepatitis B, or Hepatitis C infections.
5. History of recurrent Clostridium difficile infection or FMT in the past 6-months.
6. History of other active gastrointestinal conditions such as irritable bowel syndrome, microscopic colitis, celiac disease, short gut syndrome, colostomy, colectomy, gastrointestinal fistulae or strictures, chronic parasitic infections, diverticulitis etc.
7. Known history of bile acid diarrhea
8. Compromised immune system (e.g. primary immune disorders or clinical immunosuppression due to a medical condition or medication e.g. taking oral prednisone >20 mg a day or prednisone-equivalent)
9. History of active cancer and/or ongoing chemotherapy (superficial non-metastatic cancers and maintenance chemotherapy are permitted).
10. History of use of an investigational drug within 90 days prior to the screening visit.
11. History of significant uncontrolled systemic disease that in the opinion of the study investigator could interfere with study participation and/or objectives.
12. Life expectancy of < 1 year.
13. In the opinion of investigator, subject for any reason, should be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 58 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patients in remission after administering 12 weeks of PRIM-DJ2727 capsules will be measured by partial Mayo score ≤ 3 | 9 months

SECONDARY OUTCOMES:
Quality of life will be characterized by health-related quality of life score. | 9 months
Subject-reported score in Hospital Anxiety and Depression Scale | 9 months
  After administering 12 weeks of PRIM-DJ2727

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided